CLINICAL TRIAL: NCT05695755
Title: Postural Tachycardia Syndrome and Vasovagal Syncope in Relation to Serum Electrolytes and Adrenal Insufficiency Among Adults Attending the Main Assiut University Hospital
Brief Title: Postural Tachycardia Syndrome and Vasovagal Syncope in Relation to Serum Electrolytes and Adrenal Insufficiency
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hossam Mostafa Abdelraheem, Doctor, Assiut University
Other Study IDs: PoTS and adrenal insufficiency
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: POTS - Postural Orthostatic Tachycardia Syndrome
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Caves

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ECHO, Serum electrolytes — echocardiography, serum electrolytes and cortisol level for all patients

SUMMARY:
The present study aims to:

1. Estimate the prevalence of Postural Tachycardia Syndrome and vasovagal syncope among adults patients attend the Internal Medicine Clinic and ICU in period from 11/2022 to 10/2023
2. Detect of causes and the relationship between POTS and vasovagal syncope and serum electrolytes, and serum cortisol.

DETAILED DESCRIPTION:
Postural Orthostatic Tachycardia Syndrome (POTS) is a common, although not so well-known variant of cardiovascular autonomic disorder characterized by an excessive heart rate increase on standing, symptoms of orthostatic intolerance and maybe syncope.

The most common complaints are dizziness, weakness, rapid heartbeat and palpitation on standing. Moreover, patients often report physical deconditioning and reduced exercise capacity as well as headache, brain fog, dyspnea, gastrointestinal disorders and musculoskeletal pain.

The etiology of POTS is largely unknown and three main hypotheses include an autoimmune disorder, abnormally increased sympathetic activity and catecholamine excess and sympathetic denervation leading to central hypervolemia and reflex tachycardia. The diagnostic criteria of POTS in this study is increasing hear rate from supine position to active standing by > 30 beat per minute and positive poor mans man tilt table test.

On the other hand, Vasovagal Reflex Syncope is the most frequent cause of transient loss of consciousness . The vasovagal reaction consists of vasodilatation and a heart rate decrease. During prolonged standing, this reaction is triggered by a reduction of the central blood volume because of pooling in the lower body veins, sometimes combined with other provocative factors . Patients with reflex syncope may suffer from recurrent loss of consciousness. Most of those patients also experience frequent presyncope, which can be just as incapacitating as syncope itself. Vasovagal syncope is usually not a dangerous condition, because episodes are self-limiting. However, the quality of life of patients with recurrences can be seriously affected . The rapid loss of consciousness and the possibility of trauma tax the patients sense of physical control and self-esteem.

ELIGIBILITY:
Inclusion Criteria:

1. Patient Above 18 years.
2. Patient fulfilling diagnostic criteria of POTS increase heart rate from supine position to active standing by > 30 beat per minute within 10 minutes and positive poor mans man tilt table test.
3. Patient with History of vasovagal syncope

Exclusion Criteria:

1. Age Below 18 Yrs old
2. patient with specific cardiac diseases
3. Patient with Neurologic disorders
4. patients on drugs that affect vasomotor tone of blood vessels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with inclusion criteria attending Internal Medicine Department, The Main Assiut University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Estimate the prevalence of Postural Tachycardia Syndrome and vasovagal syncope | 11/2022 to 10/2023
  Estimate the prevalence of Postural Tachycardia Syndrome and vasovagal syncope among adults patients attend the Internal Medicine Clinic and IC Detect of causes and the relationship between POTS and vasovagal syncope and serum electrolytes, and serum cortisol.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Freeman R, Wieling W, Axelrod FB, Benditt DG, Benarroch E, Biaggioni I, Cheshire WP, Chelimsky T, Cortelli P, Gibbons CH, Goldstein DS, Hainsworth R, Hilz MJ, Jacob G, Kaufmann H, Jordan J, Lipsitz LA, Levine BD, Low PA, Mathias C, Raj SR, Robertson D, Sandroni P, Schatz IJ, Schondorf R, Stewart JM, van Dijk JG. Consensus statement on the definition of orthostatic hypotension, neurally mediated syncope and the postural tachycardia syndrome. Auton Neurosci. 2011 Apr 26;161(1-2):46-8. doi: 10.1016/j.autneu.2011.02.004. Epub 2011 Mar 9. No abstract available. PMID 21393070